CLINICAL TRIAL: NCT03410823
Title: Community Ambulation Project (CAP) Ancillary Study - PUSH Plus Protein Pilot Study
Brief Title: PUSH Plus Protein Pilot for Hip Fracture Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the extended COVID-19 shutdown, the study was terminated early with a smaller sample size of 12 included in the analyses
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Denise Orwig, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HP-00075086; R37AG009901 (NIH)
Record Dates: First submitted 2017-12-07; First posted 2018-01-25 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Hip Fracture
Keywords: hip fracture; exercise; protein
MeSH Terms: conditions — Hip Fractures; Motor Activity | interventions — Proteins; Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PUSH Plus Protein and Nutrition (Experimental): Participants will be given a whey-based protein supplement containing 27.6g of protein daily for 16 weeks and receive the PUSH intervention. PUSH is a specific multi-component intervention based on improving specific precursors to community ambulation. The intervention addresses endurance with continuous upright exercise for 20 min.; function by improving fast walking, standing from a chair, and stair negotiation; muscle performance by exercising to enhance lower extremity strength; and balance by performing unilateral activities and activities with decreased base of support. Participants receive 32 visits of approximately 60 minutes in duration from a study PT. Participants will receive two visits a week, on non-consecutive days, for 16 weeks. Visits take place in the participant's place of residence. Participants also receive the nutritional intervention for the duration of the 16-week study.
  Interventions: Behavioral: PUSH; Dietary Supplement: Protein; Dietary Supplement: Nutrition

INTERVENTIONS:
Behavioral: PUSH — Strength components of the muscle performance intervention are performed using a portable progressive resistive exercise device (Shuttle® MiniPress, Contemporary Design Company, P.O. Box 5089, Glacier, Washington 98244). Muscle performance focuses on bilateral hip extensors, hip abductors, knee extensors, and plantar flexors. Balance and strength are addressed with additional exercises performed while standing. The endurance intervention begins with 2-3 minutes of continuous upper and lower extremity active range of motion (AROM) with the participant sitting in order to increase the participants' heart rate (HR) or exertion closer to the target zone. The participant is then asked to walk on level surfaces and/or up and down steps to keep the HR within the training zone for 20 minutes.
Dietary Supplement: Protein — Participants will receive a whey-based protein supplement in the form of a powder containing 27.6g of protein. This dose induces maximum muscle protein synthesis post-exercise. Participants will mix the supplement in 8 oz of water (or other beverage) or soft food (e.g., yogurt, soup) and consume immediately following each exercise session with the study PT. On days when they do not have a physical therapy visit with the study PT, participants will be instructed to take the supplement at the meal time closest to the time of scheduled PT visits to maintain regular daily dosing schedule.
Dietary Supplement: Nutrition — Participants receive 2000 IU vitamin D3, 600 mg calcium, and a multivitamin daily for the duration of the study. Nutritional counseling is also provided. Participants are screened at baseline to assess nutritional risk using the Mini Nutritional Assessment-Short Form and contacted by a registered dietician (RD) within 7 days of baseline testing Those who score ≤7 (malnourished) and participants with baseline serum albumin 2.5-3.5 g/dl receive a visit from an RD with follow-up a week later. Participants who score 8-11 (at risk of malnutrition) and have serum albumin level >3.5 g/dl receive a phone call from the RD and may receive an in-person visit if warranted. Those screening in the normal range (12-14) and have serum albumin level >3.5 g/dl receive a phone call from the RD. Weight is monitored every 4 weeks. Those who lose 2% or more body weight receive a call from the RD. Those who lose 5% or more body weight between baseline and follow-up may be referred to an RD.

SUMMARY:
Hip fracture is a common problem among older individuals. The goal of current standard of care after hip fracture is to achieve independent, household ambulation 2-3 months after surgery, yet decreased functional ability typically persists well beyond three months and many patients never resume independent ambulation outside the home. Previous research has established that one must be able to walk at least 300 meters (~330 yards) within 6 minutes to re-establish routine interactions in the community, such as going to the store or to church. In part, this is based on the average distance from handicapped parking spaces into most facilities. Activity and exercise are believed to be of benefit for reducing disability in older adults, yet the majority of older adults does not participate in regular exercise and is not active. This is especially true for older adults following hip fracture after they complete the usual rehabilitation program.

This research study is being done to test a 16-week, multi-part exercise intervention for hip fracture patients that will be supervised by specially trained physical therapists (PTs). The exercise intervention uses a novel machine to provide strength and endurance training in the home. This has been shown in smaller studies to be safe and effective at increasing strength. The purpose of this small pilot study is to test whether adding a protein supplement to the exercise intervention leads to more improvements in a person's ability to walk in their own home and in the local community. With this knowledge, investigators hope to help a greater number of hip fracture patients enjoy a more complete recovery and improved overall health.

In addition to providing important information on adherence, feasibility, and safety, this pilot study of hip fracture patients has the unique advantage of being able to compare data to two recently completed studies where participants received the PUSH intervention without protein supplementation.

DETAILED DESCRIPTION:
A pilot study including 20 older adults who have experienced a hip fracture will be carried out with participants receiving a specific multi-component intervention with protein supplementation (PUSH Plus Protein). Study activities for participants meeting eligibility criteria will take place after post-acute rehabilitation ends, up to 26 weeks after admission to the hospital for hip fracture. Patients age 60 and older who have had surgical repair for hip fracture will be identified in study hospitals or by self-referral and evaluated for eligibility. Following consent to participate, eligible participants will undergo a comprehensive baseline assessment. Participants completing the entire baseline assessment will be eligible to receive the intervention. All participants will receive the PUSH Plus Protein intervention. The follow-up assessment will occur after the intervention is completed, approximately 16 weeks after baseline testing. The primary endpoint will be measured using the Six-Minute Walk Test (SMWT).

Participants in this pilot will receive the same specific multi-component 16-week intervention, PUSH, as participants in the multi-site randomized controlled trial, "Improving Community Ambulation after Hip Fracture (CAP)" (NCT01783704). The purpose of this study is to test whether adding a protein supplement to the PUSH intervention (PUSH Plus Protein) leads to greater improvement in a person's ability to walk in their own home and in the local community compared to the PUSH intervention alone; therefore, data in this pilot study will be compared to data from participants in the CAP study across the three sites who received the PUSH intervention alone (n=105). The working hypothesis is that PUSH Plus Protein will lead to greater improvements in ability to walk in the community compared to PUSH.

Investigators will also compare the effect of PUSH Plus Protein intervention to PUSH intervention alone on secondary outcomes in the CAP study believed to be precursors to community ambulation as shown in Aim 2 below.

Investigators can also compare participants in the pilot study to participants who received PUSH alone in the ancillary study to CAP, "Mechanistic Pathways to Community Ambulation (CAP-MP)" (n=19) to examine whether PUSH Plus Protein has an impact on the mechanistic factors on the pathway to recovery of ambulatory ability after hip fracture (Aim 3).

Aim 1. To test whether PUSH Plus Protein intervention improves community ambulation (as measured by distance walked in six minutes) compared to PUSH intervention alone (from CAP parent study) at the end of 16 weeks.

Aim 2. To assess the effects of PUSH Plus Protein on precursors to community ambulation compared to the PUSH intervention alone (CAP study). To determine the effects of PUSH Plus Protein intervention, compared to PUSH, on several other outcomes in CAP including activities of daily living (ADLs), quality of life, lower-extremity physical performance, increase of ≥ 50 meters in distance walked in six minutes, cognitive status, and nutritional status.

Aim 3. To determine the effects of PUSH Plus Protein intervention on the mechanistic factors compared to PUSH intervention alone (CAP-MP ancillary study). To determine if, at the end of the 16 week intervention, participants in the PUSH Plus Protein intervention, compared to PUSH alone, have: a) greater muscle volume and attenuation (i.e., reduced intra-muscular fat) of the thigh; b) greater lower extremity strength; c) better gait parameters; d) greater bone mineral density and bone strength; e) more bone formation and less bone resorption; and f) lower levels of circulating inflammatory cytokines.

Aim 4. To determine safety and tolerability of delivering the PUSH Plus Protein intervention to hip fracture patients. This pilot study will be used to estimate the sample size requirements for a more definitive study.

ELIGIBILITY:
Inclusion Criteria:

* Closed fracture of proximal femur
* Age 60 or older at time of baseline testing
* Minimal trauma fracture
* Non-pathologic fracture
* Surgical fixation of fracture
* Living in the community at time of fracture
* Ambulating without human assistance 2 months prior to fracture
* Unable to walk 300 m or more in 6 minutes without human assistance at time of baseline testing

Exclusion Criteria:

* Not English speaking
* Does not live within reasonable distance of the clinical center
* End stage renal disease on dialysis
* Recent myocardial infarction
* Uncompensated congestive heart failure
* Lower extremity amputation
* Symptoms of angina pectoris
* Chest pain or shortness of breath (including from severe COPD)
* Participant plans to move out of area or otherwise be unavailable during the 16-week intervention period
* Participation in another clinical trial
* Not community-residing (e.g., resident of a skilled nursing facility) at time of baseline testing
* Not fully weight-bearing on fractured leg or non-fractured leg at time of baseline testing
* Calculated creatinine clearance < 15 ml/min
* Serum albumin < 2.5 g/dl
* Hemoglobin < 9 g/dl
* Receiving physical therapy for the hip fracture in the hospital or inpatient rehabilitation facility at time of baseline testing
* Severely diminished lower extremity sensation or ulceration
* Uncontrolled hypertension
* Chronic kidney disease
* Severe liver disease (e.g., hepatitis, fatty liver disease, cirrhosis)
* Poorly controlled and/or insulin-dependent diabetes
* Known dairy allergy
* Denied medical clearance by appropriate medical provider
* Clinical site clinician thinks participant is not a good candidate for study (e.g., not likely to survive study period)
* Cognitive impairment (3MS score <73)
* Development of chest pain or substantial shortness of breath or ambulating with severe pain during baseline SMWT
* Participant walks less than 4 meters in 40 seconds (<0.1 m/sec) during baseline SMWT
* Baseline testing not done by 26 weeks post admission for hip fracture
* Final sign-off from study clinician and/or principal investigator is incomplete
* Incomplete baseline data
* Unable to contact participant
* Participant is unable to provide her/his own informed consent
* Participant refuses the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Magaziner, PhD, MSHyg, Study Chair — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Baltimore, Maryland
  - University of Maryland - St. Joseph Medical Center, Towson, Maryland

REFERENCES:
- [Background] Sallinen J, Pakarinen A, Fogelholm M, Alen M, Volek JS, Kraemer WJ, Hakkinen K. Dietary intake, serum hormones, muscle mass and strength during strength training in 49 - 73-year-old men. Int J Sports Med. 2007 Dec;28(12):1070-6. doi: 10.1055/s-2007-965003. Epub 2007 May 11. PMID 17497592
- [Background] Sallinen J, Pakarinen A, Fogelholm M, Sillanpaa E, Alen M, Volek JS, Kraemer WJ, Hakkinen K. Serum basal hormone concentrations and muscle mass in aging women: effects of strength training and diet. Int J Sport Nutr Exerc Metab. 2006 Jun;16(3):316-31. doi: 10.1123/ijsnem.16.3.316. PMID 16948487
- [Background] Chesley A, MacDougall JD, Tarnopolsky MA, Atkinson SA, Smith K. Changes in human muscle protein synthesis after resistance exercise. J Appl Physiol (1985). 1992 Oct;73(4):1383-8. doi: 10.1152/jappl.1992.73.4.1383. PMID 1280254
- [Background] Phillips SM, Tipton KD, Aarsland A, Wolf SE, Wolfe RR. Mixed muscle protein synthesis and breakdown after resistance exercise in humans. Am J Physiol. 1997 Jul;273(1 Pt 1):E99-107. doi: 10.1152/ajpendo.1997.273.1.E99. PMID 9252485
- [Background] Wolfe RR. Skeletal muscle protein metabolism and resistance exercise. J Nutr. 2006 Feb;136(2):525S-528S. doi: 10.1093/jn/136.2.525S. PMID 16424140
- [Background] Borsheim E, Tipton KD, Wolf SE, Wolfe RR. Essential amino acids and muscle protein recovery from resistance exercise. Am J Physiol Endocrinol Metab. 2002 Oct;283(4):E648-57. doi: 10.1152/ajpendo.00466.2001. PMID 12217881
- [Background] Rasmussen BB, Tipton KD, Miller SL, Wolf SE, Wolfe RR. An oral essential amino acid-carbohydrate supplement enhances muscle protein anabolism after resistance exercise. J Appl Physiol (1985). 2000 Feb;88(2):386-92. doi: 10.1152/jappl.2000.88.2.386. PMID 10658002
- [Background] Esmarck B, Andersen JL, Olsen S, Richter EA, Mizuno M, Kjaer M. Timing of postexercise protein intake is important for muscle hypertrophy with resistance training in elderly humans. J Physiol. 2001 Aug 15;535(Pt 1):301-11. doi: 10.1111/j.1469-7793.2001.00301.x. PMID 11507179
- [Background] Norton LE, Layman DK. Leucine regulates translation initiation of protein synthesis in skeletal muscle after exercise. J Nutr. 2006 Feb;136(2):533S-537S. doi: 10.1093/jn/136.2.533S. PMID 16424142
- [Background] Jackman SR, Witard OC, Jeukendrup AE, Tipton KD. Branched-chain amino acid ingestion can ameliorate soreness from eccentric exercise. Med Sci Sports Exerc. 2010 May;42(5):962-70. doi: 10.1249/MSS.0b013e3181c1b798. PMID 19997002
- [Background] Matsumoto K, Koba T, Hamada K, Sakurai M, Higuchi T, Miyata H. Branched-chain amino acid supplementation attenuates muscle soreness, muscle damage and inflammation during an intensive training program. J Sports Med Phys Fitness. 2009 Dec;49(4):424-31. PMID 20087302
- [Background] Verdijk LB, Jonkers RA, Gleeson BG, Beelen M, Meijer K, Savelberg HH, Wodzig WK, Dendale P, van Loon LJ. Protein supplementation before and after exercise does not further augment skeletal muscle hypertrophy after resistance training in elderly men. Am J Clin Nutr. 2009 Feb;89(2):608-16. doi: 10.3945/ajcn.2008.26626. Epub 2008 Dec 23. PMID 19106243
- [Background] Campbell WW, Leidy HJ. Dietary protein and resistance training effects on muscle and body composition in older persons. J Am Coll Nutr. 2007 Dec;26(6):696S-703S. doi: 10.1080/07315724.2007.10719650. PMID 18187436
- [Background] Ponzer S, Tidermark J, Brismar K, Soderqvist A, Cederholm T. Nutritional status, insulin-like growth factor-1 and quality of life in elderly women with hip fractures. Clin Nutr. 1999 Aug;18(4):241-6. doi: 10.1016/s0261-5614(99)80076-4. PMID 10578024
- [Background] Lumbers M, New SA, Gibson S, Murphy MC. Nutritional status in elderly female hip fracture patients: comparison with an age-matched home living group attending day centres. Br J Nutr. 2001 Jun;85(6):733-40. doi: 10.1079/bjn2001350. PMID 11430778
- [Background] Conigrave AD, Brown EM, Rizzoli R. Dietary protein and bone health: roles of amino acid-sensing receptors in the control of calcium metabolism and bone homeostasis. Annu Rev Nutr. 2008;28:131-55. doi: 10.1146/annurev.nutr.28.061807.155328. PMID 18466091
- [Background] Darling AL, Millward DJ, Torgerson DJ, Hewitt CE, Lanham-New SA. Dietary protein and bone health: a systematic review and meta-analysis. Am J Clin Nutr. 2009 Dec;90(6):1674-92. doi: 10.3945/ajcn.2009.27799. Epub 2009 Nov 4. PMID 19889822
- [Background] Tkatch L, Rapin CH, Rizzoli R, Slosman D, Nydegger V, Vasey H, Bonjour JP. Benefits of oral protein supplementation in elderly patients with fracture of the proximal femur. J Am Coll Nutr. 1992 Oct;11(5):519-25. doi: 10.1080/07315724.1992.10718256. PMID 1452950
- [Background] Schurch MA, Rizzoli R, Slosman D, Vadas L, Vergnaud P, Bonjour JP. Protein supplements increase serum insulin-like growth factor-I levels and attenuate proximal femur bone loss in patients with recent hip fracture. A randomized, double-blind, placebo-controlled trial. Ann Intern Med. 1998 May 15;128(10):801-9. doi: 10.7326/0003-4819-128-10-199805150-00002. PMID 9599191
- [Background] Cuthbertson D, Smith K, Babraj J, Leese G, Waddell T, Atherton P, Wackerhage H, Taylor PM, Rennie MJ. Anabolic signaling deficits underlie amino acid resistance of wasting, aging muscle. FASEB J. 2005 Mar;19(3):422-4. doi: 10.1096/fj.04-2640fje. Epub 2004 Dec 13. PMID 15596483
- [Background] Ryan AS, Dobrovolny CL, Smith GV, Silver KH, Macko RF. Hemiparetic muscle atrophy and increased intramuscular fat in stroke patients. Arch Phys Med Rehabil. 2002 Dec;83(12):1703-7. doi: 10.1053/apmr.2002.36399. PMID 12474173
- [Background] Goodpaster BH, Carlson CL, Visser M, Kelley DE, Scherzinger A, Harris TB, Stamm E, Newman AB. Attenuation of skeletal muscle and strength in the elderly: The Health ABC Study. J Appl Physiol (1985). 2001 Jun;90(6):2157-65. doi: 10.1152/jappl.2001.90.6.2157. PMID 11356778
- [Background] Mourtada FA, Beck TJ, Hauser DL, Ruff CB, Bao G. Curved beam model of the proximal femur for estimating stress using dual-energy X-ray absorptiometry derived structural geometry. J Orthop Res. 1996 May;14(3):483-92. doi: 10.1002/jor.1100140319. PMID 8676262
- [Background] Beck TJ, Ruff CB, Warden KE, Scott WW Jr, Rao GU. Predicting femoral neck strength from bone mineral data. A structural approach. Invest Radiol. 1990 Jan;25(1):6-18. doi: 10.1097/00004424-199001000-00004. PMID 2298552
- [Background] Guigoz Y, Vellas B, Garry PJ. Assessing the nutritional status of the elderly: The Mini Nutritional Assessment as part of the geriatric evaluation. Nutr Rev. 1996 Jan;54(1 Pt 2):S59-65. doi: 10.1111/j.1753-4887.1996.tb03793.x. No abstract available. PMID 8919685
- [Background] Wells JL, Dumbrell AC. Nutrition and aging: assessment and treatment of compromised nutritional status in frail elderly patients. Clin Interv Aging. 2006;1(1):67-79. doi: 10.2147/ciia.2006.1.1.67. PMID 18047259
- [Background] Vellas B, Guigoz Y, Garry PJ, Nourhashemi F, Bennahum D, Lauque S, Albarede JL. The Mini Nutritional Assessment (MNA) and its use in grading the nutritional state of elderly patients. Nutrition. 1999 Feb;15(2):116-22. doi: 10.1016/s0899-9007(98)00171-3. PMID 9990575
- [Background] Sato T, Matsuyama Y. Marginal structural models as a tool for standardization. Epidemiology. 2003 Nov;14(6):680-6. doi: 10.1097/01.EDE.0000081989.82616.7d. PMID 14569183
- [Background] Rubin DB. Estimating causal effects from large data sets using propensity scores. Ann Intern Med. 1997 Oct 15;127(8 Pt 2):757-63. doi: 10.7326/0003-4819-127-8_part_2-199710151-00064. PMID 9382394
- [Background] Perera S, Mody SH, Woodman RC, Studenski SA. Meaningful change and responsiveness in common physical performance measures in older adults. J Am Geriatr Soc. 2006 May;54(5):743-9. doi: 10.1111/j.1532-5415.2006.00701.x. PMID 16696738
- [Background] Cohen J. Statistical power analysis for the behavioral sciences. 2nd ed. Hillsdale, NJ: Lawrence Erlbaum Associates, 1988.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were evaluated for eligibility in 3 phases out to 26 weeks post admission in 7 area hospitals (2019-2020). We screened 440 hip fracture patients at Phase 1 and 143 (32%) were eligible based on medical chart review. After Phase 2 and 3 screening, 20 (20%) people were enrolled and screened at Phase 2. Of those who consented, 3 were found to be ineligible at Phase 3, 2 refused, 1 was not able to have baseline testing within timeframe, and 14 participants completed baseline testing
Pre-assignment Details: Of those who consented, 3 were found to be ineligible at Phase 3, 2 refused, 1 was not able to have baseline testing within timeframe, and 14 participants completed baseline testing
Groups:
- PUSH Plus Protein and Nutrition: This PUSH+Protein pilot study had the unique advantage of being able to compare data to the recently completed recruitment and intervention-matched study (CAP: n=35)) and its ancillary study (CP-MP: n=20) [Sep 2013 - Oct 2017 (ClinicalTrials.gov Identifier: NCT01783704)] conducted at 1 of 3 clinical sites where participants received the PUSH intervention without protein supplementation.
  PUSH+Protein pilot study (2019-2020) utilized the same recruitment and screening procedures, inclusion and exclusion criteria, PUSH intervention, and vitamins and nutritional supplements, as the CAP study. Participants received a micro-filtrated unflavored whey protein isolate powder (gluten and lactose free) from True Nutrition (Vista, CA) with 27.6g of protein in a scoop taken daily. Participants mixed the protein powder in 8 oz. of water (or other cold beverage) or soft food (e.g., yogurt) and consumed it immediately following each exercise session with the study physical therapist. On days when they did not have a visit with the study physical therapist, participants were instructed to take the supplement at the mealtime closest to the time of scheduled PT visits to maintain a regular daily dosing schedule. 20 people were enrolled and 14 completed baseline testing and initiated in-home PUSH sessions.
Period: Overall Study
Arm/Group | PUSH Plus Protein and Nutrition
Started | 14
Completed | 9
Not Completed | 5
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Withdraw due to COVID-19 shutdown | 2

BASELINE CHARACTERISTICS:
Population: Participants were hip fracture patients 60 years of age and older with surgical repair enrolled within 26 weeks post admission who were living in the community at the time the time of baseline testing.
Groups:
- PUSH Plus Protein and Nutrition: Participants received a whey-based protein powder containing 27.6g of protein per scoop taken daily for 16 weeks. Participants will mix the supplement in 8 oz of water (or other beverage) or soft food (e.g., yogurt, soup) and consume immediately following each exercise session with the study PT and at same time on other days of the week. Participants also received the PUSH intervention delivered in the home by a study PT [2 times/wk for 32 visits (approx. 60 minutes per visit)] over 16 weeks. Strength components of the muscle performance intervention were performed using a portable progressive resistive exercise device (Shuttle® MiniPress, Contemporary Design Company, P.O. Box 5089, Glacier, Washington 98244). Muscle performance focused on bilateral hip extensors, hip abductors, knee extensors, and plantar flexors. Balance and strength were addressed with additional exercises performed while standing. The endurance intervention began with 2-3 minutes of continuous upper and lower extremity active range of motion (AROM) with the participant sitting in order to increase the participants' heart rate (HR) or exertion closer to the target zone. The participant was then asked to walk on level surfaces and/or up and down steps to keep the HR within the training zone for 20 minutes. Participants also received the nutritional counseling and daily supplements (600 mg calcium, 2000 IU vitamin D, and multivitamin) for the duration of the 16-week study.
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 82.07 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Fracture type [Count of Participants; unit: Participants]
  Femoral neck | 4
  Pertrochanteric | 10
Comorbidities [Mean (Standard Deviation); unit: number of comorbidities] | 5.07 (3.54)
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.2 (6.09)
3MS [Mean (Standard Deviation); unit: units on a scale] — The Modified Mini-Mental State (3MS) is a widely used assessment capturing cognitive status. The 3MS test has a score range of 1-100 with higher scores indicating better cognitive function. It can be used to monitor cognitive change over time.
  units on a scale | 89.93 (9.08)
6-minute walk test distance [Mean (Standard Deviation); unit: meters] — The Six-Minute Walk Test (SMWT) will be used to obtain a continuous measure of total distance walked in six minutes.
  meters | 180.12 (48.10)
SPPB [Mean (Standard Deviation); unit: units on a scale] — The SPPB evaluates lower extremity performance in older persons based on timed short distance walk, repeated chair stands, and a set of balance tests. Each of the tasks is assigned a score ranging from 0 to 4, with 4 indicating the highest level of performance and 0 an inability to complete the test. A higher score indicates better performance. The scores range from 0-12.
  units on a scale | 5.0 (2.51)
MNA-SF [Mean (Standard Deviation); unit: score on a scale] — Nutritional status will be assessed using the Mini Nutritional Assessment-Short Form (MNA®-SF), a validated and widely used malnutrition screening tool. We are using a modified version of the MNA®, approved by the scale's developer (the Nestlé company), to facilitate use as an interviewer-administered tool in a research setting. Scores range from 0 to 14; participants scoring ≤7 will be considered malnourished; those scoring 8-11 will be considered to be at risk of malnutrition; and those scoring 12-14 will be considered to have normal nutritional status.
  score on a scale | 9.07 (2.30)

OUTCOME MEASURES:

1. Primary Outcome: Distance Walked in Six Minutes
Description: The Six-Minute Walk Test (SMWT) will be used to obtain a continuous measure of total distance walked in six minutes. The SMWT is highly correlated with workloads, heart rate, oxygen saturation, and dyspnea responses when compared to bicycle ergometry and treadmill exercise tests in older persons. It has been performed by elderly, frail and severely compromised participants who cannot perform standard maximal treadmill or cycle ergometry exercise tests.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 9
meters | 179.84 (60.14)

2. Secondary Outcome: Cognitive Function (3MS)
Description: The Modified Mini-Mental State (3MS) is a widely used assessment of cognitive status. The 3MS test has a score range of 1-100 with higher scores indicating better cognitive function.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 9
units on a scale | 92.78 (8.26)

3. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: The SPPB evaluates lower extremity performance in older persons based on timed short distance walk, repeated chair stands, and a set of balance tests. Each of the tasks is assigned a score ranging from 0 to 4, with 4 indicating the highest level of performance and 0 an inability to complete the test. A higher score indicates better performance. The scores range from 0-12.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 9
units on a scale | 5.44 (2.24)

4. Secondary Outcome: Activities of Daily Living (ADLs)
Description: We will measure ADLs using a modified version of the Pepper Assessment Tool for Disability (PAT-D) with two modifications. First, two items (walking a quarter mile and walking across a small room) were added to address perceived gaps in the original PAT-D scale. This modification is consistent with the version used in the Lifestyle Interventions and Independence for Elders study. Second, two items (walking several blocks and lifting heavy objects) were deleted to avoid duplication with other items in the scale, resulting in a 19-item scale with higher scores indicating worse function. There are 3 subscales: Basic (score range 1-5), instrumental (score range 1-5), and functional (score range 1-5) (formerly mobility subscale).
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 9
score on a scale
  Basic Subscale | 1.41 (0.54)
  Functional Subscale: number analyzed (Participants) | 8
  Functional Subscale | 1.98 (0.72)
  Instrumental Subscale: number analyzed (Participants) | 6
  Instrumental Subscale | 1.08 (0.20)

5. Secondary Outcome: Quality of Life (SF-36)
Description: We will use an interviewer-administered version of the SF-36 ( 36-Item Short Form Health Survey) , a health survey that assesses quality of life in eight subscales [physical function, social function, role-physical, role-emotional, bodily pain, mental health, general health, and vitality]. The SF-36 has been validated as a generic measure of quality of life in many different populations, including patient and non-patient samples. Each of the subscales has a score range of 0-100 and we only used 4 subscales (role-physical, vitality, social functioning, and role-emotional). Higher scores indicate higher quality of life through less disability across the 8 domains.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 9
score on a scale
  Role Physical | 50.0 (41.46)
  Vitality | 56.67 (14.14)
  Social Functioning | 86.11 (22.92)
  Role Emotional | 74.07 (43.39)

6. Secondary Outcome: Nutritional Status
Description: Nutritional status will be assessed using the Mini Nutritional Assessment-Short Form (MNA®-SF), a validated and widely used malnutrition screening tool. We are using a modified version of the MNA®, approved by the scale's developer (the Nestlé company), to facilitate use as an interviewer-administered tool in a research setting. Scores range from 0 to 14; participants scoring ≤7 will be considered malnourished; those scoring 8-11 will be considered to be at risk of malnutrition; and those scoring 12-14 will be considered to have normal nutritional status.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 9
score on a scale | 12.33 (2.29)

7. Secondary Outcome: Body Composition- Done Density
Description: Bone density will be estimated using dual-energy x-ray absorptiometry (DXA) (GE LUNAR, Madison, WI). DXA calculates BMD (g.cm2) at the Total Hip and Femoral Neck regions and values are provided in the report produced by the DXA machine.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 8
g/cm2
  Total Hip BMD: number analyzed (Participants) | 7
  Total Hip BMD | .72 (.10)
  Femoral neck BMD: number analyzed (Participants) | 7
  Femoral neck BMD | .71 (.09)

8. Secondary Outcome: Muscle Composition
Description: A single computed tomography (CT) scan at the mid-thigh region using a Siemens Somatom Sensation 64 Scanner (Fairfield, CT) was used to assess muscle area, high density lean tissue, and low density lean tissue area (IMAT),all on the fracture and non fracture sides. The CT was analyzed using MIPAV (NIH Image Analysis Visualization Progam, v.7.0).
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 9
cm2
  High density muscle -fractured side | 46.83 (11.90)
  High density muscle- non fractured side | 55.65 (15.43)
  Low density muscle-fractured side | 26.04 (8.45)
  Low density muscle-non fractured side | 25.73 (8.30)

9. Secondary Outcome: Power
Description: A Biodex System 3 PRO dynamometer will measure strength per unit of time (power) for bilateral knee flexion-extension. Power is measured in Watts (W). Testing will utilize standardized positioning and joint motion excursions. Subjects performed three repetitions and the values across the three trials were averaged for the power value.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: W
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 6
W
  Knee extension-fracture side | 20.21 (7.71)
  Knee extension-non fracture side | 24.51 (8.70)
  Knee flexion-fracture side | 12.28 (2.69)
  Knee flexion-non fracture side | 15.84 (2.52)

10. Secondary Outcome: Strength
Description: A Biodex System 3 PRO dynamometer will measure max power over the entire range of motion (strength) for bilateral knee flexion-extension. Strength is measured in Newton-meters (Nm). Testing will utilize standardized positioning and joint motion excursions. Subjects performed three repetitions and the values across the three trials were averaged for the strength value.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 6
Nm
  Knee extension-fracture side | .34 (.13)
  Knee extension-non fracture side | .40 (.14)
  Knee flexion-fracture side | .21 (.05)
  Knee flexion-non fracture side | .27 (.04)

11. Secondary Outcome: Bone Turnover Markers - Bone Formation
Description: Bone formation (serum aminoterminal propeptide of type 1 procollagen; P1NP (ug/l)) will be assessed.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: ug/l
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 8
ug/l | 86.69 (52.02)

12. Secondary Outcome: Bone Turnover Markers - Bone Resorption
Description: Bone resorption (serum cross-linked C-telopeptides of type I collagen; CTx-I (ng/mL)) will be assessed.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 8
ng/ml | .50 (.19)

13. Secondary Outcome: Hormones
Description: Insulin Growth Factor (IGF-1) will be measured by ELISA.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 8
ng/ml | 127.05 (31.94)

14. Secondary Outcome: Inflammatory Cytokines
Description: a) interleukin-6 (IL-6) and b) soluble TNF- α receptor 1 (sTNF- αR1). Both cytokines were measured in serum by ELISA (R&D Systems Inc., Minneapolis, MN) and expressed at pg/ml levels.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 8
pg/mL
  TNF-alpha R1 | 1685.88 (510.15)
  IL-6 | 4.81 (2.34)

15. Secondary Outcome: GAITrite Distance
Description: A GAITrite instrumented walkway system will measure spatial and temporal gait parameters. Subjects will walk at their safest fast and natural speeds. Distance (spatial) variables will include step length (cm).Each participant completed two trials of each condition with a short rest period between trials for a total of four trials (i.e., 2 trials × 2 conditions). For each condition, values were averaged over the two trials. Walking aids were permitted only when the participant needed the aid to walk independently.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 8
cm
  Normal Walk distance | 723.11 (33.39)
  Fast Walk distance | 699.39 (38.24)

16. Secondary Outcome: GAITrite Velocity
Description: A GAITrite instrumented walkway system will measure spatial and temporal gait parameters. Subjects will walk at their safest fast and natural speeds. Time (temporal) variables include walking speed. Each participant completed two trials of each condition with a short rest period between trials for a total of four trials (i.e., 2 trials × 2 conditions). For each condition, values were averaged over the two trials. Walking aids were permitted only when the participant needed the aid to walk independently.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 8
cm/sec
  Normal walk speed | 58.99 (13.04)
  Fast walk speed | 81.01 (22.88)

17. Secondary Outcome: Four-Square Step Test
Description: The Four Square Step Test (FSST) is used to assess dynamic stability and the ability of the subject to step over low objects forward, sideways, and backward. The FSST may be an effective and valid tool for measuring dynamic balance and the subject's fall risk.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 4
seconds | 10.32 (14.24)

18. Secondary Outcome: Cognitive Function (Trail Making Test (Trails A & B))
Description: The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning. It is sensitive to detecting cognitive impairment associated with dementia.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 7
seconds
  Trails A | 96.33 (82.59)
  Trails B | 185.0 (79.09)

19. Secondary Outcome: Body Composition- Lean Body Mass
Description: Muscle and lean mass will be estimated using dual-energy x-ray absorptiometry (DXA) (GE LUNAR, Madison, WI). DXA calculates lean muscle mass (kg) from the total body scan and values are provided in the report produced by the DXA machine. The coefficient of variation of these measurements in our previous studies for lean mass was 1.3%.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 8
kg | 40.16 (57.65)

20. Other Pre Specified Outcome: Adherence With PUSH Intervention
Description: PTs will submit a visit form for each of the 32 visits that records date of visit; start and end time of the visit; reason for missed visit; what activities were performed; and whether activities were performed as prescribed. For the PUSH group, we will also obtain information about the intensity of each activity at initiation of the intervention and every four weeks during the intervention period. Logs completed by PTs will record the detail of each designated activity during intervention sessions as well as any precautions or modifications to activities. Reasons for protocol variations will be noted in the PT log books.
Time Frame: 16 weeks
Population: Participants eligible to receive the 16-week intervention.
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 12
number of visits | 25.33 (11.74)

21. Other Pre Specified Outcome: Adherence With Protein Supplement
Description: We will monitor adherence to the protein supplement by weighing the container(s) of protein powder every 4 weeks during the 16-week intervention period to derive an average daily consumption.
Time Frame: 16 weeks
Population: Participants who were eligible to receive the entire 16-week intervention.
Measure: Mean (Full Range); unit: grams per day
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 12
grams per day | 26.42 [25.81 to 27.2]

22. Secondary Outcome: Muscle Composition-attenuation
Description: A single computed tomography (CT) scan at the mid-thigh region using a Siemens Somatom Sensation 64 Scanner (Fairfield, CT) was used to assess muscle attenuation in Hounsfield units (HU) on the fracture and non fracture sides. The CT was analyzed using MIPAV (NIH Image Analysis Visualization Progam, v.7.0). HUs are used by radiologists to interpret CT images and differentiate between tissues and fluids. Muscle attenuation is a measure of muscle density that correlates with the amount of fat in the muscles. Lower HU values indicate higher levels of intramuscular fat. Therefore, decreased muscle attenuation has been linked to reduced strength and performance. A normal HU for low-density muscle is 0-34.
Time Frame: 16 weeks
Population: Participants who initiated the intervention and had a 16-week follow-up visit.
Measure: Mean (Standard Deviation); unit: HU
Arm/Group | PUSH Plus Protein and Nutrition
Number analyzed (Participants) | 9
HU
  Muscle Attenuation (HU)- fracture side | 14.45 (8.07)
  Muscle Attenuation (HU)-non fracture side | 19.85 (7.28)

ADVERSE EVENTS:
Time Frame: The requirements for reporting RAEs began when the participant provided informed consent and ended 30 days after the participant's involvement (up to 16 weeks) in the study was completed.
Description: In this study, reportable AEs (RAEs) are defined as serious adverse events (SAEs), AEs that have potential implications for participant safety, unexpected AEs, and injury that occurs while a participant is under the supervision of study-related personnel. These RAEs require individual event reporting. Classification of SAEs and AEs related to severity, expectedness and relatedness does not differ the standard definitions.
Arm/Group | PUSH Plus Protein and Nutrition
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PUSH Plus Protein and Nutrition (N=12)
Pneumonia (Infections and infestations) | 1 (1) — Hospitalized for cardiopulmonary and abdominal concerns and the outcome was fatal.
Cholecystitis (Infections and infestations) | 1 (1) — Hospitalized for infected gall bladder duct

LIMITATIONS AND CAVEATS:
The PUSH + Protein Pilot study was originally powered for 30 participants. However, due to the extended COVID-19 shutdown, the study was terminated early with a smaller sample size of 12 included in the analyses. As a result, we did not analyze all of the secondary outcomes originally planned. Since the pilot study provided important feasibility data for using protein supplement in older hip fracture patients, data analyses were conducted on the primary outcome and a few key secondary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT03410823/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT03410823/SAP_001.pdf